CLINICAL TRIAL: NCT03231748
Title: Clearance of Inflammatory Cytokines in Patients With Septic Acute Kidney Injury During Renal Replacement Therapy Using the EMIC®2 Filter
Brief Title: Clearance of Inflammatory Cytokines During Renal Replacement Therapy Using the EMIC®2 Filter
Acronym: ClicAKI
Status: Completed | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS ID: 196972
Record Dates: First submitted 2017-07-10; First posted 2017-07-27 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Acute Renal Failure
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will be conducted in patients with sepsis and acute kidney injury needing renal replacement therapy.

The aim is to investigate whether continuous renal replacement therapy with the EMIC®2 filter leads to removal of pro-inflammatory middle molecular weight cytokines from the blood.

DETAILED DESCRIPTION:
In patients with acute kidney injury (AKI) and sepsis requiring renal replacement therapy, the investigators aim to determine whether continuous veno-venous haemodialysis with an EMiC®2 filter leads to clearance of the following mediators Interleukin (IL) -1 alpha, IL-1 beta, IL-2, IL- 4, IL-6, IL-8, IL-10, Tissue necrosis factor alpha (TNF-α), vascular endothelial growth factor (VEGF), Interferon gamma, Monocyte chemotactic protein-1 and epidermal growth factor.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (≥18 years) in the Critical Care Unit with AKI and sepsis
* clinical decision that citrate based continuous veno-venous haemodialysis (CVVHD) is necessary

Exclusion Criteria:

* lack of consent
* pre-existing dialysis dependent renal failure
* life expectancy <24 hours
* patients with haemoglobin <7g/dL (unless transfused for clinical reasons)
* need for extracorporeal membrane oxygenation (ECMO)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with sepsis and acute kidney injury who require renal replacement therapy.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Removal of inflammatory mediators | 48 hours
  Clearance of the following mediators Interleukin (IL) -1 alpha, IL-1 beta, IL-2, IL- 4, IL-6, IL-8, IL-10, Tissue necrosis factor alpha (TNF-α), vascular endothelial growth factor (VEGF), Interferon gamma, Monocyte chemotactic protein-1 and epidermal growth factor

SECONDARY OUTCOMES:
Adsorption of inflammatory mediators | 48 hours
  Adsorption of IL-1 alpha, IL-1 beta, IL-2, IL- 4, IL-6, IL-8, IL-10, Tissue necrosis factor alpha (TNF-α), vascular endothelial growth factor (VEGF), Interferon gamma, Monocyte chemotactic protein-1 and epidermal growth factor

CONTACTS AND LOCATIONS:
Overall Officials: Marlies Ostermann, PhD, Study Director — Guy's & St Thomas Hospital London
Locations (1):
- Guy's & St Thomas Hospital, London, United Kingdom

REFERENCES:
- [Derived] Lumlertgul N, Hall A, Camporota L, Crichton S, Ostermann M. Clearance of inflammatory cytokines in patients with septic acute kidney injury during renal replacement therapy using the EMiC2 filter (Clic-AKI study). Crit Care. 2021 Jan 28;25(1):39. doi: 10.1186/s13054-021-03476-x. PMID 33509215